CLINICAL TRIAL: NCT05060406
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of LY06006 in Postmenopausal Women With Osteoporosis at High Risk for Fracture
Brief Title: A Study to Evaluate the Efficacy and Safety of LY06006 in Postmenopausal Women With Osteoporosis at High Risk for Fracture
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shang Dong Boan Biotechnology Co., Ltd (Co-sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY06006/CT-CHN-302
Record Dates: First submitted 2021-04-20; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: It is a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY06006 60mg (Experimental): injection
  Interventions:
  Drug: LY06006 Injection； Dietary Supplement: Elemental Calcium； Dietary Supplement: Vitamin D
  Interventions: Drug: LY06006
- Placebo (Placebo Comparator): injection
  Interventions:
  Drug: Placebo； Dietary Supplement: Elemental Calcium； Dietary Supplement: Vitamin D
  Interventions: Drug: LY06006

INTERVENTIONS:
Drug: LY06006 — 60 mg/1 ml, once every 6 months administered subcutaneously, two injections in total
  Other Names: recombinant human monoclonal anti-RANKL antibody injection

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled phase III clinical study will be conducted to evaluate the efficacy and safety of LY06006 in the treatment of postmenopausal women with osteoporosis at high risk for fracture, as well as an exploratory population pharmacokinetic analysis of LY06006.

DETAILED DESCRIPTION:
It is a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial.

Primary Objective:

To evaluate the efficacy of LY06006 in the treatment of postmenopausal women with osteoporosis at high risk for fracture.

Secondary Objectives:

To evaluate the safety of LY06006. To evaluate the immunogenicity of LY06006. Population pharmacokinetic analysis of LY06006.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal woman, ages ≥50 to ≤85 years.≥3 years postmenopausal, which can be≥3 years of spontaneous amenorrhea or ≥3 years post-surgical bilateral oophorectomy. If < 60 years of age and had hysterectomy but ovarian retention, require follicle stimulating hormone (FSH) levels ≥40U/L.

   Exclusion Criteria:
2. Low BMD (BMD absolute value consistent with a T-score≤-2.5 and >-4.0 at either the lumbar spine or total hip). The BMD equivalents by T-score thresholds for each DXA scanner manufacturer are provided below.
3. Have at least one of the following risk factors:

   1. history of fragility fracture
   2. parental history of hip fracture
   3. low body weight (BMI≤19kg/m2)
   4. elderly (age≥65y)
   5. current smoker
4. Voluntarily signed written informed consent

Exclusion criteria

1. Bone/metabolic disease:

   1. Any metabolic bone disease, e.g., osteomalacia or osteogenesis imperfecta,
   2. Paget's disease
   3. Cushing's disease
   4. Hyperprolactinemia
   5. Hypopituitarism
   6. Acromegaly
   7. Current hyperparathyroidism or hypoparathyroidism by medical record.
   8. Current hyperthyroidism or hypothyroidism (allowed if having normal hormone level on thyroid hormone replacement therapy or 5.5μIU/mL<thyroid-stimulating hormone (TSH) level≤10.0μIU/mL, but the serum thyroxine (T4) is within the normal range.
   9. Malabsorption syndrome or any gastrointestinal disorders associated with malabsorption, for example Crohn's Disease and chronic pancreatitis.
   10. Hypocalcemia or hypercalcemia, or serum albumin corrected blood calcium level is not within the normal range of the laboratory;
   11. Vitamin D deficiency: 25 hydroxy vitamin D (25OHD) level <20 ng/mL. (allowed 200,000 units of vitamin D2 injection (trade name: Futai®) once during the screening period, and re-test the 25OHD level once. Those with 25OHD level ≥20 ng/mL can be included
   12. Others such as rheumatoid arthritis, gout, multiple myeloma and so on.
2. Subjects with a history of greater than 2 vertebral fractures.
3. Malignancy within the 5 years before enrollment (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical or breast ductal carcinoma in situ).
4. Severe renal disease, creatinine clearance <30mL/min
5. Liver or biliary diseases:

   1. Cirrhosis of the liver;
   2. Biliary tract abnormalities (except asymptomatic gallstones);
   3. Positive Hepatitis C virus (HCV) antibody;
   4. Positive hepatitis B surface antigen (HBsAg) test with the peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) titer test ≥1×103 copies/mL (if positive HBsAg with the peripheral blood HBV DNA titer test <1× 103 copies/mL, the subject is eligible for selection if the investigator believes that the subject is in a stable phase of chronic hepatitis B and will not increase the risk of the subject,;
   5. Alkaline phosphatase <lower limit of normal (LLN); alkaline phosphatase or total bilirubin ≥ 1.5 times the upper limit of normal (ULN); serum aspartate aminotransferase (AST) ≥ 2.0×ULN; serum alanine Acid aminotransferase (ALT) ≥2.0×ULN;
6. Oral/Dental Diseases

   1. Prior history or current evidence of osteomyelitis or osteonecrosis of the jaw.
   2. Active dental or jaw condition which requires oral surgery.
   3. Planned invasive dental procedure.
   4. Non-healed dental or oral surgery.
7. DXA measurements:

   1. Less than two lumbar vertebrae evaluable for DXA measurements.
   2. Height, weight, or girth that could preclude accurate DXA measurements.
8. Administration of the following medications:

   1. RANKL inhibitor, fluoride or strontium salt or intravenous bisphosphonate within the past 5 years;
   2. Oral bisphosphonates, allowed if patients had the following conditions :

      * Cumulative use> 3 months but <3 years: ≥ 6 months before the last medication was taken from the screening visit;
      * Cumulative use ≤3 months;
   3. parathyroid hormone (PTH) or parathyroid hormone analogs (PTHa) within 6 weeks before screening, such as teriparatide; anabolic hormones or testosterone; glucocorticoids (equivalent to> 5 mg/day strength Pine> 10 days); systemic hormone replacement therapy; selective estrogen receptor modulators (SERMs), such as raloxifene; tibolone; calcitonin; active vitamin D and its analogs; other bone active drugs including anticonvulsants (except benzodiazepines) and heparin; long-term systemic use of ketoconazole, androgens, corticotropin, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, Gonadotropin releasing hormone agonist;
9. Positive human immunodeficiency virus (HIV) antibody.
10. Self-reported alcohol or drug abuse [defined as drinking an average of 14 units or more of alcoholic beverages per week in the 3 months before screening (1 unit = 350 mL of beer, or 45 mL of liquor, or 150 mL of wine)]
11. Known allergy to the treatment drugs used in the research protocol, including allergy to the test drugs
12. Have received any other experimental drug treatment or prior participation in another interventional clinical trial within 3 months before screening
13. Other severe acute or chronic diseases, psychiatric disorder or abnormal laboratory tests, etc., in the opinion of the investigator, not suitable for participating in this research.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal woman
Enrollment: 448 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) at the Lumbar Spine | Baseline and Month 12
  Percent Change From Baseline in Bone Mineral Density (BMD) at the Lumbar Spine at Month 12

SECONDARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) at the Lumbar Spine | Baseline and Month 6
  Percent Change From Baseline in BMD at the Lumbar Spine at Month 6
Percent Changes in total hip BMD | Baseline,Month 6 and Month 12
  Percent Changes in total hip BMD from baseline at 6 and 12 months of treatment
Percent Changes in femoral neck BMD | Baseline,Month 6 and Month 12
  Percent Changes in femoral neck BMD from baseline at 6 and 12 months of treatment
Percent Changes in trochanteric BMD | Baseline,Month 6 and Month 12
  Percent Changes in trochanteric BMD from baseline at 6 and 12 months of treatment
Percent Change in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) From Baseline | Baseline, Month 1, Month 6 and Month 12
  Percent Change From Baseline in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) From Baseline at Month 1, Month 6, and Month 12
Percent Change in Serum Procollagen Type I N Propeptideserum (s-PINP) From Baseline | Baseline, Month 1, Month 6 and Month 12
  Percent Change From Baseline in Serum Procollagen Type I N Propeptideserum (s-PINP) From Baseline at Month 1, Month 6, and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlin Zhang, doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No